CLINICAL TRIAL: NCT00577759
Title: Community and Clinician Partnership for Prevention
Acronym: C2P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00004061; HHSA290200710014
Record Dates: First submitted 2007-12-13; First posted 2007-12-20 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2012-10

CONDITIONS: Physical Activity; Dietary Habits; Tobacco Use Cessation
Keywords: Quality assurance, health care; primary health care; community health services; referral and consultation; exercise; diet; tobacco
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Intervention (Experimental): Direct referral to community organizations, with support for practices to do so. These include the North Carolina Tobacco Quitline, public health department dietitians, and the YMCA.
  Interventions: Other: Active Intervention
- Passive Intervention (Experimental): Provision of information about community organizations to patients as above.
  Interventions: Other: Passive Intervention
- Usual Care (Placebo Comparator): Usual care
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Active Intervention — Quality improvement activities, including monthly teleconferences and chart audit with feedback, to help practices refer to community resources
  Arms: Active Intervention
Other: Passive Intervention — Provision of tools to help with referrals to community resources
  Arms: Passive Intervention
Other: No intervention — No intervention
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the impact of strategies to develop and foster the relationship between primary care practices and community resources to address specific unhealthy behaviors (tobacco use, poor nutrition, and lack of physical activity).

DETAILED DESCRIPTION:
Tobacco use, poor diet, and lack of physical activity are associated with the leading causes of significant morbidity and mortality, including coronary heart disease, hypertension, cancer, stroke, diabetes, and respiratory dysfunction. One solution to decreasing unhealthy behaviors would be to better integrate primary care providers with community resources, including community and public health organizations that already have the capacity and expertise to deliver effective interventions. This project is a randomized trial to evaluate different practice-level interventions to link practices to community resources to decrease unhealthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine and family practices in Durham and Orange counties, North Carolina

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The number of referrals from the practices to the community resources | 6 months

SECONDARY OUTCOMES:
Number of referrals received by each resource | 6 months
The proportion of patients with unhealthy behaviors who were referred from the practices to community resources | 6 months
Practice attitudes and practice regarding referral to community resources | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Kemper, MD, MPH, MS, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States